CLINICAL TRIAL: NCT05740670
Title: An Open-label Clinical Trial to Investigate the Safety and Efficacy of a Bone Broth Diet on Weight Loss in Obese Adults
Brief Title: The Safety and Efficacy of a Bone Broth Diet on Weight Loss in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veyl Ventures LLC (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22VVCFB01
Record Dates: First submitted 2023-01-26; First posted 2023-02-23 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Weight Loss
Keywords: Safety and efficacy; Weight loss; Obesity; Bone broth
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dr. Kellyann's Bone Broth (Experimental): During the bone broth phases, each week will be separated into 'fasting days' and 'feeding days'. There will be 2 non-consecutive fasting days and 5 feeding days per week. On fasting days, participants will be instructed to consume 1 packet of bone broth every 2 hours, for a total of 7 packets/day. On feeding days, participants will consume 3 meals/day, made up of 'Yes' foods portioned according to instructions provided in the Bone Broth Diet Quick Reference Guide and 1 packet of bone broth, twice a day, as snacks between meals. If a bone broth serving is missed participants are instructed to consume the serving as soon as they remember. Participants will be advised not to exceed 7servings of bone broth on fasting days and 2 servings on feeding days. During the maintenance phase, participants will not consume any bone broth.
  Interventions: Other: Dr. Kellyann's Bone Broth

INTERVENTIONS:
Other: Dr. Kellyann's Bone Broth — Participants will have two bone broth phases, each three weeks in length. Bone broth phases will be separated by a one-week maintenance phase. A one-week maintenance phase will also occur after the second bone broth phase. Each week of a broth phase will consist of five feeding days and five fasting days. On feeding days, participants will consume one packet of bone broth, twice each day, as snacks between meals. On fasting days, participants will consume one packet of bone broth every two hours for a total of seven packets each day.

SUMMARY:
The primary objective of this study is to investigate the safety and efficacy of a bone broth diet on weight loss in obese adults. The change in weight and body mass index (BMI) following the bone broth diet will be measured from baseline at Days 22 and 50. Additionally, the safety and tolerability of the bone broth diet will be measured by the occurrence of post-emergent adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the age of 35-65 years, inclusive, at screening
2. BMI between 30.0 and 39.9 kg/m2
3. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle and agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence and agrees to use contraception if planning on becoming sexually active
4. Agrees to maintain current lifestyle habits as much as possible throughout the study depending on your ability to maintain the following: medications, supplements, and sleep
5. Motivated to comply with dietary and fasting guidelines as assessed by the Motivation Questionnaire at screening (see Appendix 16.2)
6. Self-reported stable body weight for the past three months defined as not having gained or lost more than 5 kg of body weight throughout the three months prior to screening
7. Willingness and ability to complete questionnaires, records, and diaries associated with the study, adhere to dietary/fasting guidelines, read the Revised Bone Broth Diet book (chapters 1-5), and to complete all clinic visits
8. Provided voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance to the investigational product's ingredients
3. Metal implants or other physical characteristics/limitations that may affect DEXA scan results, as assessed by the QI
4. Participation within the last three months in any weight loss or diet programs from baseline
5. Current or history of eating disorders, as assessed by the QI
6. Obesity-induced by metabolic or endocrinologic disorders (ex. acromegaly, hypothalamic obesity), as assessed by the QI
7. Current or history of significant diseases of the gastrointestinal tract, as assessed by the QI
8. Gastric bypass surgery or other surgeries to induce weight loss
9. History of gout and have had a flare up within past 12 months
10. Chronic inflammatory diseases, as assessed by the QI
11. Type I or Type II diabetes (HbA1c ≥6.5%)
12. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
13. Current unstable diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
14. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
15. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
16. Current use of any prescribed or over-the counter medications and/or supplements that may affect body weight or metabolism, as assessed by the QI (See Sections 7.3.1and 7.3.2)
17. Regular use of tobacco products within 6 months of baseline and during the study period, as assessed by the QI
18. Alcohol intake average of >2 standard drinks per day. Occasional users must agree to wash out and abstain during the study period, as assessed by the QI
19. Alcohol or drug abuse within the last 12 months
20. Use of medical cannabinoid products
21. Chronic use of cannabinoid products (>2 times/week). Occasional users must agree to wash out and abstain during the study period
22. Clinically significant abnormal laboratory results at screening, as assessed by the QI
23. Blood donation 30 days prior to baseline, during the study, or a planned donation within 30 days of the end of study
24. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
25. Individuals who are unable to give informed consent
26. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
The change in weight from baseline at Days 22 and 50 following the bone broth diet. | baseline, day 22, day 50
The change in body mass index (BMI) from baseline at Days 22 and 50 following the bone broth diet. | baseline, day 22, day 50

SECONDARY OUTCOMES:
The change in weight from baseline at Day 28, from Day 22 at Day 28, from Day 28 at Day 50, and from Day 50 at Day 56 following the bone broth diet. | baseline, day 22, day 28, day 50, day 56
The change in body mass index (BMI) from baseline at Day 28, from Day 22 at Day 28, from Day 28 at Day 50, and from Day 50 at Day 56 following the bone broth diet. | baseline, day 22, day 28, day 50, day 56
The change in android/gynoid fat ratio from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
  The change in android/gynoid fat ratio from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet as assessed by DEXA measurements.
The change in fat mass (percent or grams) from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
  The change in fat mass from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet as assessed by DEXA measurements.
The change in muscle mass (percent or grams) from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
  The change in muscle mass from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet as assessed by DEXA measurements.
The change in waist circumference from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
The change in sagittal abdominal diameter (SAD) from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
The change in hip circumference from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
The change in arm circumference from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
The change in thigh circumference from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
The change in waist-to-hip ratio from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
The change in blood glucose levels from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
The change in triglyceride levels from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
The change in total cholesterol levels from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
The change in high-density lipoprotein cholesterol (HDL-C) levels from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
The change in non-high-density lipoprotein cholesterol (non-HDL-C) levels from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
The change in low-density lipoprotein cholesterol (LDL-C) levels from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
The change in triglyceride to high-density cholesterol ratio from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
The change in low-density cholesterol to high-density cholesterol ratio from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
The change in quality of life from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. | baseline, day 22, day 28, day 50
  The change in quality of life is assessed by the Modified Short Form (SF)-36 Quality of Life Questionnaire from baseline at Days 22, 28, and 50 and from Day 28 at Day 50 following the bone broth diet. The SF-36 measures nine scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, mental health, and reported health transition. The scores range from 0 to 100 where higher scores indicate a better state of health.

OTHER OUTCOMES:
The incidence of pre-emergent and post-emergent adverse events (AE). | baseline to day 50
Blood pressure (BP) at screening, baseline, day 22, day 28, and day 50 following the bone broth diet. | screening, baseline, day 22, day 28, day 50
Heart rate (HR) at screening, baseline, day 22, day 28, and day 50 following the bone broth diet. | screening, baseline, day 22, day 28, day 50
Serum aspartate aminotransferase (AST) measurement at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Serum alanine aminotransferase (ALT) measurement at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Serum alkaline phosphatase (ALP) measurement at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Serum total bilirubin measurement at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Creatinine measurement at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Measurement of electrolytes (sodium, potassium, chloride) at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Measurement of uric acid at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Estimated glomerular filtration rate (eGFR) at screening day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
White blood cell count (WBC) at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
White blood cell count (WBC) with differentials at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
  WBC with differentials (neutrophils, lymphocytes, monocytes, eosinophils, basophils) will be measured in the serum at screening, day 22, and day 50.
Red blood cell count (RBC) at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Hemoglobin at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Hematocrit at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Platelet count at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Immature granulocytes at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Nucleated red blood cells (RBC) at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Red blood cell (RBC) indices at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
  RBC indices include mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), and red blood cell distribution width (RDW).
Urine color and appearance at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Urinalysis-chemistry for urinary glucose at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Urinalysis-chemistry for urinary ketones at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Urinalysis-chemistry for urinary specific gravity at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Urinalysis-chemistry for blood at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Urinalysis-chemistry for urinary pH at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Urinalysis-chemistry for urinary proteins at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Urinalysis-chemistry for urinary nitrite at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50
Urinalysis-chemistry for urinary leukocytes at screening, day 22, and day 50 following the bone broth diet. | screening, day 22, day 50

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada